CLINICAL TRIAL: NCT05545761
Title: The Effect of Music Therapy on Sleep Quality and Depression in Menopausal Women: A Randomized Controlled Study
Brief Title: The Effect of Music Therapy on Sleep Quality and Depression in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meryem Vural Şahin (Other)
Responsible Party: Sponsor-Investigator, Meryem Vural Şahin, PHD Student, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: meryemvrlshn00000000001
Record Dates: First submitted 2022-09-07; First posted 2022-09-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2022-12

CONDITIONS: Menopause
Keywords: music therapy; depression; sleep quality
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): music will be played to the intervention group. They will be asked to listen to the Hüseyni makam for at least 15 minutes at 11.00 in the morning, 5 times a week for 5 weeks, and to listen to the Zirgüle makam for at least 15 minutes at 20.00 on the same day.
  Interventions: Other: music therapy
- control group (No Intervention): group that does not listen to music and is not interfered with

INTERVENTIONS:
Other: music therapy — Feedback will be received via WhatsApp that the participants have listened to the maqam conveyed to them.Before applying music therapy in the experimental group, they will be asked to fill out the questionnaires.At the end of the music therapy application, the questionnaires made at the beginning will be applied to the experimental group again.No application will be made to the control group, and data collection forms will be applied twice with an interval of 4 weeks.
  Arms: intervention group

SUMMARY:
About one-third of women experience no or mild symptoms during their menopausal life, while another third experience moderate symptoms, while the remaining one-third may experience severe symptoms.

It is stated that hormone therapy, one of the pharmacological methods, is accepted as an effective and standard method in the management of menopausal symptoms, including sleep disorders and depression, despite its side effects. However, due to the health risks associated with hormone therapy, it is stated that many women do not want to use this treatment option and turn to complementary and alternative medicine to alleviate menopausal symptoms. It is stated that physical, mental and psychological problems of women can be treated with non-pharmacological methods such as relaxation, breathing exercises, touch therapy, and music therapy as a complementary and alternative medicine approach in the world and in Turkey.

It is stated that the healing effect of music has been known among societies since ancient times. Today, with technological developments, it is stated that music does not only rest the soul, but also has a cognitively stimulating effect and a motivating effect in cases where verbal communication cannot be performed. When the national and international literature is examined, there are many studies on non-pharmacological methods for menopausal symptoms, while the effect of music therapy on depression in menopausal women was examined in only one study in Turkey. However, no study was found in which the music therapy method was used for both depression and sleep quality in menopausal women.

For this reason, the aim of the study was to determine the effect of music therapy, which is a non-pharmacological method, on sleep quality and depression in menopausal women.

DETAILED DESCRIPTION:
According to WHO, the menopausal period is not a pathological process, but is expressed as one of the biological stages of a woman's life. The menopausal period is defined as the transition to old age, which begins with regression in ovarian functions and decreased reproductive capacity, and in time, reproductive ability ends.

Approximately one-third of women experience no symptoms or mild symptoms during the menopausal period, while the other third experience moderate symptoms, while the remaining one-third may experience severe symptoms. The symptomatology experienced in this period is characterized by a hypoestrogenic state that occurs due to regression in ovarian function in 60% to 80% of women . In addition to symptoms such as insomnia, vaginal dryness, irregular menstrual bleeding, depressed mood, irritability, headache, forgetfulness, and dizziness, vasomotor symptoms such as changes in body thermoregulation and night sweats can be observed in menopausal women as a result of insufficient secretion of sex hormones.

Sleep problems are defined as one of the important problems seen in menopausal women It is stated that hot flashes and especially night sweats seen in the menopausal period may cause sleep disorders with the slowdown in serotonin metabolism due to hypoestrogen. While sleep problems can negatively affect mood and activities of daily living in women, it has been reported that they have a wide-ranging negative impact on quality of life, mood, productivity and physical health, especially in women with severe sleep problems. It is stated that sleep disorders do not only affect the quality of life in women in the menopausal period, but may cause social burdens by jeopardizing their lives and health in the long run.

It is stated that depression affects approximately 350 million people worldwide and is a global burden. It is stated that depression is seen twice as often in women as in men, and that the risk of depression may increase during periods when women experience hormonal changes such as puberty, pregnancy, and transition to menopause.It is stated that the menopausal period, in which hormonal changes are experienced intensively, is not associated with psychiatric diseases alone, but the risk of its occurrence increases, especially in women in the perimenopausal period, even if there is no previous history of depressive disorder.

It is stated that hormone therapy, one of the pharmacological methods, is accepted as an effective and standard method in the management of menopausal symptoms, including sleep disorders and depression, despite its side effects. However, due to the health risks associated with hormone therapy, it is stated that many women do not want to use this treatment option and turn to complementary and alternative medicine to alleviate menopausal symptoms. It is stated that physical, mental and psychological problems of women can be treated with non-pharmacological methods such as relaxation, breathing exercises, touch therapy, and music therapy as a complementary and alternative medicine approach in the world and in Turkey.

It is stated that the healing effect of music has been known among societies since ancient times. Today, with technological developments, it is stated that music does not only rest the soul, but also has a cognitively stimulating effect and a motivating effect in cases where verbal communication cannot be performed. The importance of music therapy and its relationship with treatment was emphasized by Florence Nightingale in the early 1800s, and it was used as a therapeutic approach, accepted the power of the use of appropriate music in the healing of patients and defined music therapy as a part of the healing process Lafcı in 2018 found that music therapy had positive effects on sleep and anxiety in women with breast cancer. Kavurmacı in 2019 found that music therapy positively affects sleep quality in their study with students. It is stated that music has a therapeutic effect on mental illnesses such as depression by regulating the stress response of the hypothalamus-pituitary-adrenal axis. According to the meta-analysis results in which music therapy studies applied to patients with digestive tumors were examined, it was determined that the sleep quality could be improved and the level of depression could be reduced in those who received music therapy. It was found that music therapy had a significant effect on sleep quality and depression in patients who applied to the psychiatry outpatient clinic due to insomnia in Iran. Koçak in 2022 found that music therapy positively affects depression in menopausal women.

When the national and international literature is examined, there are many studies on non-pharmacological methods for menopausal symptoms, while the effect of music therapy on depression in menopausal women was examined in only one study in Turkey. However, no study was found in which the music therapy method was used for both depression and sleep quality in menopausal women.

Based on this argument, a study was planned to examine the effect of music therapy on sleep quality and depression in menopausal women.

Material and Method The research will be carried out with menopausal women who applied to Çayyolu No. 1 FHC between August 2022 and December 2022. The research was designed as a randomized controlled experimental study. The sample of the study was G-Power 3.1.7; By comparing the sleep quality scores between the groups, it was planned to have 35 cases in the experimental and control groups.Sampling will be done by dividing the menopausal women who apply to the FHC, who meet the inclusion criteria, into the experimental and control groups at a rate of 1/1. Considering the risk of data loss in both groups, 20% more cases will be taken.

Since the variables to be examined in our study are depression and sleep quality, the type of music to be used will be zirgüle makam and Hüseyni makam. When the effects of authorities on the human spirit are examined; It is stated that while the zirgüle maqam gives people sleep, the huseyni maqam gives people comfort . A WhatsApp group will be created with the experimental group. The links of the authority that will be played via Whatsapp will be sent.They will be asked to listen to the Hüseyni makam for at least 15 minutes at 11.00 in the morning, 5 times a week for 5 weeks, and to listen to the Zirgüle makam for at least 15 minutes at 20.00 on the same day. Feedback will be received via WhatsApp that the participants have listened to the maqam conveyed to them.Before applying music therapy in the experimental group, they will be asked to fill out the questionnaires.At the end of the music therapy application, the questionnaires made at the beginning will be applied to the experimental group again.No application will be made to the control group, and data collection forms will be applied twice with an interval of 4 weeks.

Data Collection Tools

1. Sociodemographic Information Form The first 9 questions question the participant's sociodemographic characteristics such as age, weight, height, occupation, educational status, and the next 10 questions consist of questions prepared to determine the obstetrical characteristics.While the next question was asked to detect the presence of chronic disease in the person, the last two questions were asked to detect the presence of cancer and depression.The sociodemographic information form consists of 21 questions in total.
2. Beck Depression Inventory In the study, Beck Depression Inventory will be used to evaluate the presence and severity of depression symptoms.The inventory was developed by Beck (1961) in order to express the degree of depression objectively through numbers.The Turkish adaptation of the inventory was made by Hisli (1988).For each of the 21 items that make up the inventory, there are four self-evaluation statements rated from zero to three, ranking the severity of the symptom from least to greatest.The lowest score that can be obtained from the inventory is 0 and the highest score is 63.The high total score indicates the high level of depression or its severity.In addition, a cut-off point of 17 is recommended for catching clinical depression.
3. Menopause Symptoms Rating Scale The scale was developed by the Berlin Center for Epidemiology and Health Research The validity and reliability study in Turkey was conducted by Metintaş in 2009.The 11-item Likert-type scale including menopausal complaints consists of 3 sub-dimensions.Somatic complaints sub-dimension; Items 1, 2, 3, 11, psychological complaints sub-dimension; 4th, 5th, 6th, 7th items and urogenital complaints sub-dimension; It includes items 8, 9, 10. For each item; 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe and the minimum score that can be taken from the scale is 0, and the maximum score is 44.An increase in the total score obtained from the scale indicates that both the severity of the complaints experienced and the quality of life are negatively affected.
4. Pittsburg Sleep Quality Scale (PUKÖ) It was developed by Buysse in 1989, and its validity and reliability study in Turkey was performed by Ağargün in 1996. PUKÖ consists of a total of 24 questions. 19 of the questions are self-evaluation questions, 5 of them are answered by the spouse or relative.Question 19 is not taken into account in scoring. PUKO; It consists of seven items evaluating subjective sleep quality, sleep delay, sleep duration, sleep efficiency, sleep disturbance, use of sleeping pills, and impairment in daytime work. Each component is evaluated with a score between 0-3.The scale total score is between 0-21. A PUKÖ total score of 5 and above indicates poor sleep quality.Its diagnostic sensitivity is 89.6% and its specificity is 86.5%. It takes 5-10 minutes to complete the scale

Evaluation of Data The data will be analyzed in SPSS program. Student's t test will be used for two independent group variables with normal distribution, Mann Whitney U test for data that is not normally distributed, and chi-square test for categorical variables

ELIGIBILITY:
Inclusion Criteria:

* Menopausal
* PSQI average score of 5 and above
* No hearing problem
* Not taking HRT at the time of the study or in the past year
* There was no diagnosis of a psychiatric disease during the study.

Exclusion Criteria:

Having communication problems, Receiving HRT treatment during the study or in the last year, Not attending music therapy sessions,

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — menopausal
Enrollment: 70 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PUKI) | 5 weeks after the start of music therapy
  The maximum and minimum total scores that can be obtained from the Pittsburgh sleep quality index (PUKI) scale range from 0 to 21. Sleep quality will be defined as poor in women who score 5 or more on this scale.
Beck Depression Scale | 5 weeks after the start of music therapy
  While the maximum score to be obtained from the Beck Depression Scale is 63, it will be accepted that the presence and severity of depression increase as the score from the scale increases. The woman who gets a maximum of 10 points will be defined as no depression.
Menopausal Symptoms Evaluation Scale | 5 weeks after the start of music therapy
  The total score that can be obtained from the Menopausal Symptoms Evaluation Scale is between 0-44. The increase in the total score obtained from the scale indicates the increase in the severity of the complaints.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - University of Health Sciences Gülhane Faculty of Health Sciences, Ankara
  - Meryem VURAL ŞAHİN, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Augoulea A, Moros M, Lykeridou A, Kaparos G, Lyberi R, Panoulis K. Psychosomatic and vasomotor symptom changes during transition to menopause. Prz Menopauzalny. 2019 Jun;18(2):110-115. doi: 10.5114/pm.2019.86835. Epub 2019 Jun 28. PMID 31485208
- [Background] Trimarco V, Rozza F, Izzo R, De Leo V, Cappelli V, Riccardi C, Di Carlo C. Effects of a new combination of nutraceuticals on postmenopausal symptoms and metabolic profile: a crossover, randomized, double-blind trial. Int J Womens Health. 2016 Oct 11;8:581-587. doi: 10.2147/IJWH.S115948. eCollection 2016. PMID 27785106
- [Background] Chen X, Wei Q, Jing R, Fan Y. Effects of music therapy on cancer-related fatigue, anxiety, and depression in patients with digestive tumors: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2021 Jun 4;100(22):e25681. doi: 10.1097/MD.0000000000025681. PMID 34087821
- [Background] Weidner K, Bittner A, Beutel M, Goeckenjan M, Brahler E, Garthus-Niegel S. The role of stress and self-efficacy in somatic and psychological symptoms during the climacteric period - Is there a specific association? Maturitas. 2020 Jun;136:1-6. doi: 10.1016/j.maturitas.2020.03.004. Epub 2020 Mar 13. PMID 32386660
- [Background] Zhang J, Shao S, Ye C, Jiang B. A Clinical Study of the Effect of Estradiol Valerate on Sleep Disorders, Negative Emotions, and Quality of Life in Perimenopausal Women. Evid Based Complement Alternat Med. 2021 Oct 16;2021:8037459. doi: 10.1155/2021/8037459. eCollection 2021. PMID 34697549
- [Background] Heinemann LA, Potthoff P, Schneider HP. International versions of the Menopause Rating Scale (MRS). Health Qual Life Outcomes. 2003 Jul 30;1:28. doi: 10.1186/1477-7525-1-28. PMID 12914663
- [Background] Mehrnoush V, Darsareh F, Roozbeh N, Ziraeie A. Efficacy of the Complementary and Alternative Therapies for the Management of Psychological Symptoms of Menopause: A Systematic Review of Randomized Controlled Trials. J Menopausal Med. 2021 Dec;27(3):115-131. doi: 10.6118/jmm.21022. PMID 34989185
- [Background] Kocak DY, Varisoglu Y. The effect of music therapy on menopausal symptoms and depression: a randomized-controlled study. Menopause. 2022 May 1;29(5):545-552. doi: 10.1097/GME.0000000000001941. PMID 35486946
- [Background] Djapardy V, Panay N. Alternative and non-hormonal treatments to symptoms of menopause. Best Pract Res Clin Obstet Gynaecol. 2022 May;81:45-60. doi: 10.1016/j.bpobgyn.2021.09.012. Epub 2021 Nov 17. PMID 34952794
- [Background] Kavurmaci M, Dayapoglu N, Tan M. Effect of Music Therapy on Sleep Quality. Altern Ther Health Med. 2020 Jul;26(4):22-26. PMID 31221932
- [Background] Hachul H, Monson C, Kozasa EH, Oliveira DS, Goto V, Afonso R, Llanas AC, Tufik S. Complementary and alternative therapies for treatment of insomnia in women in postmenopause. Climacteric. 2014 Dec;17(6):645-53. doi: 10.3109/13697137.2014.926321. Epub 2014 Jul 16. PMID 24884736
- [Background] Lafci, D. (2018). Breast cancer, sleep and music therapy. Journal of Uludag University Faculty of Medicine, 44(1), 61-64.
- [Background] Hisli, N. (1988). A study on the validity of the Beck Depression Inventory. Journal of Psychology, 6(22), 118-122
- [Background] Metintas S, Arykan I, Kalyoncu C, Ozalp S. Menopause Rating Scale as a screening tool in rural Turkey. Rural Remote Health. 2010 Jan-Mar;10(1):1230. Epub 2010 Mar 31. PMID 20356316
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Gözüyenice, E., & Başer, M. (2016). Vasomotor Complaints Experienced in Menopausal Period. Anatolian Journal of Nursing and Health Sciences, 19(4).
- [Background] Orlowski, D. D., Can, U. K., & Bagci, H. (2021). Investigation of Scientific Publications in the Field of Music Therapy in Germany (2010-2019). Motif Academy Journal of Folklore, 14(33), 266-286.
- [Background] Ocebe, D. K., Kolcu, M., & Kadriye, U. Z. U. N. (2019). Music Therapy and Elderly Health. Health Sciences University Journal of Nursing, 1(2), 112-115.
- [Background] Velioğlu, E., & Gürkan, Ö. C. (2021). Evidence-Based Complementary and Alternative Therapies in the Management of Menopausal Symptoms. Journal of Traditional and Complementary Anatolian Medicine, 3(2), 20-27.
- [Background] Zhao K, Bai ZG, Bo A, Chi I. A systematic review and meta-analysis of music therapy for the older adults with depression. Int J Geriatr Psychiatry. 2016 Nov;31(11):1188-1198. doi: 10.1002/gps.4494. Epub 2016 Apr 19. PMID 27094452
- [Background] Şahan, Ö., & Oskay, Ü. M. R. A. N. (2021). Sleep changes and management in the postmenopausal period. Journal of Health Academics, 8(4), 350-359.
- [Background] Amiri, S., Parvizi Fard, A., Khaledi-Paveh, B., Foroughi, A., Bavafa, A., Bazani, M., ... & Sadeghi, K. (2019). The effect of music therapy using Persian traditional music on insomnia. Kermanshah Medical Sciences University Journal, 23
- [Background] E. E. M. Elsabagh and E. S. Abd Allah, "Menopausal symptoms and the quality of life among pre/post-menopausal women from rural area in Zagazig city," Life Science Journal, vol. 9, no. 2, pp. 283-291, 2017.